CLINICAL TRIAL: NCT04299464
Title: A Phase II Multicenter, Randomized, Double-Blind, 12-Week Treatment, 3-Arm, Parallel-Group, Placebo-Controlled Study to Investigate the Efficacy, Safety, and Tolerability of RO7017773 in Participants Aged 15-45 Years With Autism Spectrum Disorder (ASD)
Brief Title: A 12-Week Placebo-Controlled Study to Investigate the Efficacy, Safety, and Tolerability of RO7017773 in Participants Aged 15-45 Years With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP41316; 2019-003524-20 (EudraCT Number)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo matched to RO7017773 for approximately 12 weeks.
  Interventions: Drug: Placebo
- RO7017773 Low Dose (Experimental): Participants will receive a fixed low dose of RO7017773 for approximately 12 weeks.
  Interventions: Drug: RO7017773
- RO7017773 High Dose (Experimental): Participants will receive a fixed high dose of RO7017773 for approximately 12 weeks.
  Interventions: Drug: RO7017773

INTERVENTIONS:
Drug: Placebo — Participants will receive oral placebo for approximately 12 weeks.
  Arms: Placebo
Drug: RO7017773 — Participants will receive oral RO7017773 for approximately 12 weeks.
  Arms: RO7017773 High Dose; RO7017773 Low Dose

SUMMARY:
This study will investigate the efficacy, safety, tolerability, and pharmacokinetics of RO7017773 in participants aged 15-45 years who have been diagnosed with ASD with a score of >/=50 on the Wechsler Abreviated Scale of Intelligence (WASI-II).

ELIGIBILITY:
Inclusion Criteria

* Male and female participants with Autism Spectrum Disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Wechsler Abbreviated Scale of Intelligence (WASI-II) >/= 50 at screening or within the last 12 months prior to screening
* ASD or Autism diagnosis confirmed by Autism Diagnostic Observation Schedule (ADOS-2)
* Body mass index within the range of 18.5 to 40 kg/m2
* Female Participants: is eligible if she is not pregnant, not breastfeeding, and women of childbearing potential (WOCBP), who agree to remain abstinent or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 28 days after the last dose of study drug
* Language, hearing, and vision compatible with the study measurements as judged by the Investigator
* Allowed existing treatment regimens should be stable for 8 weeks prior to screening. Investigator expects stability of these treatments and behavioral interventions for the duration of the study
* In the Investigator's opinion, able to participate and deemed appropriate for participation in the study, capable of following the study SoA and able to comply with the study restrictions
* In the Investigator's opinion, participation in the study or discontinuation of prohibited medication will not pose undue risks

Exclusion Criteria

Neurologic/Psychiatric Conditions:

* Non-verbal individuals
* Presence of chromosome 15q11.2 q13.1 duplication syndrome (Dup15q syndrome), known "syndromic" forms of ASD (confirmed per genetic results available at screening): fragile X syndrome, Prader Willi syndrome, Rett's syndrome, tuberous sclerosis, and Angelman syndrome, as well as genetic alterations strongly associated with ASD per genetic results available at screening affecting the following genes: CHD8, ANDP, SHANK3
* Medical history of alcohol and/or substance abuse/dependence in the last 12 months or positive test for drugs of abuse at screening
* Initiation of a major change in psychosocial intervention within 6 weeks prior to screening. Minor changes in ongoing treatment are not considered major changes
* Clinically significant psychiatric and/or neurological disorder that may interfere with the safety or efficacy endpoints
* Risk of suicidal behavior in the opinion of a certified clinician or as evidenced by a "yes" to questions 4 and/or 5 of Columbia-Suicide-Severity Rating Scale (C-SSRS) taken at screening and baseline with respect to the last 12 months, or any suicide attempt in the past 5 years
* Unstable epilepsy/seizure disorder within the past 6 months or changes in anticonvulsive therapy within the last 6 months

Other Conditions:

* Medical history of malignancy if not considered cured or if occurred within the last 3 years with the exception of fully excised non-melanoma skin cancers or in-situ carcinoma of the cervix that has been successfully treated
* Concomitant disease, condition or treatment which would either interfere with the conduct of the study or pose an unacceptable risk to the participant in the opinion of the Investigator Prior/Concomitant Therapy
* Use of prohibited medications or herbal remedies within 6 weeks or 5 half-lives (t1/2) prior to randomization

Prior/Concurrent Clinical Study Experience:

* Donation or loss of blood over 500 mL in adults and 250 mL in adolescents within 3 months prior to randomization
* Participation in an investigational drug study within 1 month or 5 times the t1/2 of the investigational molecule prior to randomization or participation in a study testing an investigational medical device within 1 month prior to randomization or if the device is still active Diagnostic Assessments
* Confirmed clinically significant abnormality in hematological, chemistry or coagulation laboratory parameters
* Positive test result at screening for hepatitis B surface antigen, hepatitis C virus (HCV, untreated), or human immunodeficiency virus (HIV)-1 and -2. HCV participants who have been successfully treated and who test negative for HCV RNA, may be considered eligible for entry into the study

Other Exculsions:

* Uncorrected hypokalemia or hypomagnesaemia

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (11):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Yale University / Yale-New Haven Hospital, New Haven, Connecticut
  - APG- Advanced Psychiatric Group, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Nathan Kline Institute, Orangeburg, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
- Canada (4):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Janeway Childrens Health, St. John's, Newfoundland and Labrador
  - Holland Bloorview Kids Rehabilitation Hospital, East York, Ontario
  - London Health Sciences Centre, London, Ontario
- Italy (3):
  - Ist. G. Gaslini, Genoa, Liguria
  - Istituto Scientifico Medea, Bosisio Parini (LC), Lombardy
  - P.O. Gaspare Rodolico, Catania, Sicily
- Spain (3):
  - IGAIN (Instituto Global de Atención Integral al Neurodesarrollo), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 26 investigative sites in 4 countries (United States, Canada, Spain, and Italy) from 31 March 2021 to 15 May 2024.
Pre-assignment Details: A total of 104 participants diagnosed with autism spectrum disorder (ASD) were randomized in 1:1:1 ratio to receive alogabat 20 mg, 60 mg and placebo.
Groups:
- Placebo: Participants received alogabat matching placebo, orally, once daily (QD) up to 12 weeks during the treatment period.
- Alogabat 20 mg: Participants received alogabat, 20 milligrams (mg), orally, QD up to 12 weeks during the treatment period.
- Alogabat 60 mg: Participants received alogabat, 60 mg, orally, QD up to 12 weeks during the treatment period.
Period: Overall Study
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Started | 34 | 34 | 36
Completed | 32 | 30 | 29
Not Completed | 2 | 4 | 7
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Non-compliance with Study Drug | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 3
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Placebo: Participants received alogabat matching placebo, orally, QD up to 12 weeks during the treatment period.
- Alogabat 20 mg: Participants received alogabat, 20 mg, orally, QD up to 12 weeks during the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg | Total
Number analyzed (Participants) | 34 | 34 | 36 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (8.1) | 24.8 (7.1) | 25.0 (7.5) | 25.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 25 | 26 | 27 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 6 | 23
  Not Hispanic or Latino | 22 | 28 | 29 | 79
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 3 | 7
  White | 31 | 28 | 27 | 86
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Adaptive Behavior Composite (ABC) Score of the Vineland Adaptive Behavior Scales, Third Edition (Vineland-3)
Description: Vineland-3 is a semi-structured interview that measures an individual's adaptive behavior across 3 domains: Communication, Socialization, and Daily Living skills. Each domain is composed of 3 subdomains. Subdomain raw score is based on item responses (3-point scale: 0=never present; 1=sometimes present; 2=usually present) and is calculated for each subdomain of the three main domains as the sum of the scores for each item within the subdomain. Raw scores of the 9 subdomains are used to derive Growth Scale Values (GSVs; range = 10-197). A conversion table for mapping raw scores to GSV scores is found in Appendix 3, Table B.2 in the Vineland-3 manual (Sparrow et al. 2016). GSV is a person-ability score used to track an individual's progress. Vineland-3 ABC Composite GSV score is calculated as the mean GSV score (summing the 9 GSV subdomain scores and dividing by 9; Vineland-3 ABC Composite GSV scores can range from 10-154). A higher score indicates better adaptive functioning.
Time Frame: Baseline to Week 12
Population: Efficacy population included all participants who gave informed consent, were randomized, and received at least one dose of double-blind study medication. Overall number analyzed is the number of participants with data available for analysis
Measure: Mean (80% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 32 | 27 | 28
score on a scale | 3.250 [2.011 to 4.490] | 2.819 [1.469 to 4.169] | 2.807 [1.499 to 4.115]
Statistical Analysis 1: Comparison: Placebo vs Alogabat 20 mg; Test type: Superiority; p = 0.7650, ANCOVA; Difference in Adjusted Mean = -0.432, 80% CI 2-sided [-2.291 to 1.428]
Statistical Analysis 2: Comparison: Placebo vs Alogabat 60 mg; Test type: Superiority; p = 0.7517, ANCOVA; Difference in Adjusted Mean = -0.4444, 80% CI 2-sided [-2.250 to 1.363]

2. Secondary Outcome: Number of Participants With at Least One Adverse Events (AEs)
Description: An AE is an untoward medical occurrence in a participant administered a pharmaceutical product and regardless of the causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product.
Time Frame: Up to Week 18
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 34 | 34 | 36
Participants | 24 | 22 | 22

3. Secondary Outcome: Number of Participants With at Least One Serious Adverse Events (SAEs)
Description: An AE is an untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of an investigational product, whether or not considered related to investigational product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 18
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 34 | 34 | 36
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Discontinuing Treatment Due to AEs
Description: as for outcome 2
Time Frame: Day 1 up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 34 | 34 | 36
Participants | 1 | 0 | 2

5. Secondary Outcome: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behaviour as Measured Using the Columbia-Suicide-Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, and attempts with actual/potential lethality. Categories have binary responses (yes/no) and include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here.
Time Frame: Baseline up to Week 18
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 34 | 34 | 36
Participants
  Wish to be Dead | 2 | 1 | 1
  Non-specific Active Suicidal Thoughts | 1 | 1 | 1
  Self-Injurious Behavior Without Suicidal Intent | 1 | 0 | 1

6. Secondary Outcome: Change From Baseline in Karolinska Sleepiness Scale (KSS) Score for Assessing Daytime Sleepiness
Description: The KSS measures the subjective level of sleepiness at a particular time during the day. On this scale, participants (or support persons for adolescents aged 15 to 17 years and low-functioning participants) indicate which level best reflects the psycho-physical state experienced in the last 5 minutes. The KSS is a 9-point scale (1=extremely alert, 9=very sleepy, great effort to keep awake, fighting sleep). A decrease in KSS score or negative change from baseline indicate an improvement in sleepiness.
Time Frame: Baseline (Day 1 Predose), 3-4 hours post-dose on Day 1, Predose and 3-4 hours post-dose on Days 14, 42, and 84
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 33 | 34 | 36
score on a scale
  Baseline (Day 1: Predose) | 4.97 (2.10) | 4.88 (2.28) | 4.17 (2.37)
  Change from Baseline at Day 1: 3-4 hours Post Dose: number analyzed (Participants) | 33 | 33 | 36
  Change from Baseline at Day 1: 3-4 hours Post Dose | -0.88 (2.00) | -0.58 (2.12) | 0.19 (2.20)
  Change from Baseline at Day 14: Predose: number analyzed (Participants) | 33 | 32 | 31
  Change from Baseline at Day 14: Predose | -0.03 (1.91) | -0.13 (2.12) | -0.03 (2.15)
  Change from Baseline at Day 14: 3-4 hours Post Dose: number analyzed (Participants) | 33 | 32 | 32
  Change from Baseline at Day 14: 3-4 hours Post Dose | -0.76 (1.70) | -0.84 (2.60) | 0.34 (2.72)
  Change from Baseline at Day 42: Predose: number analyzed (Participants) | 32 | 31 | 31
  Change from Baseline at Day 42: Predose | -0.50 (2.05) | -0.94 (2.66) | -0.94 (1.82)
  Change from Baseline at Day 42: 3-4 hours Post Dose: number analyzed (Participants) | 31 | 31 | 31
  Change from Baseline at Day 42: 3-4 hours Post Dose | -0.74 (1.77) | -1.00 (2.79) | -0.26 (2.34)
  Change from Baseline at Day 84: Predose: number analyzed (Participants) | 31 | 29 | 29
  Change from Baseline at Day 84: Predose | -1.52 (2.23) | -0.83 (2.65) | -0.48 (2.13)
  Change from Baseline at Day 84: 3-4 hours Post Dose: number analyzed (Participants) | 31 | 30 | 27
  Change from Baseline at Day 84: 3-4 hours Post Dose | -1.13 (2.00) | -0.83 (2.80) | -0.30 (2.45)

7. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale Score (ESS) for Assessing Daytime Sleepiness
Description: The ESS is a brief, self-administered eight-item questionnaire that measures daytime sleepiness in adults. Participants were asked to rate on a scale of 0-3 the chances that, "over the past month" and "since last visit", he/she would have dozed in eight specific situations that are commonly met in daily life (0 = would never doze and 3 = high chance of dozing). The ESS score is the sum of eight item-scores and can range from 0 to 24. A lower ESS score or a negative change from baseline score indicates an improvement in daytime sleepiness.
Time Frame: Baseline (Day 1), Days 14, 42, and 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 26 | 26 | 26
score on a scale
  Baseline (Day 1) | 5.00 (3.69) | 6.15 (4.23) | 4.54 (2.67)
  Change from Baseline at Day 14: number analyzed (Participants) | 25 | 25 | 26
  Change from Baseline at Day 14 | 0.24 (2.42) | -0.72 (3.36) | 0.73 (4.58)
  Change from Baseline at Day 42: number analyzed (Participants) | 26 | 25 | 24
  Change from Baseline at Day 42 | 0.62 (2.52) | -2.08 (4.15) | 0.50 (3.39)
  Change from Baseline at Day 84: number analyzed (Participants) | 26 | 24 | 23
  Change from Baseline at Day 84 | 0.38 (3.40) | -1.46 (4.28) | 0.26 (3.41)

8. Secondary Outcome: Change From Baseline ESS Score for Children and Adolescents (ESS-CHAD) for Assessing Daytime Sleepiness
Description: The ESS-CHAD is a brief, support person-administered eight-item questionnaire that measures daytime sleepiness in children and adolescents. Each item asked the support persons of adolescents and participants with an IQ score <70 to rate on a scale of 0-3 the chances that "Over the past month," and "since last visit", "your child" would have dozed in eight specific situations that are commonly met in daily life ( 0 to 3 where 0 = would never doze and 3 = high chance of dozing). The ESS score is the sum of eight item scores and can range from 0 to 24. A lower ESS score or negative change from baseline score indicates an improvement in daytime sleepiness.
Time Frame: Baseline (Day 1), Days 14, 42, 63, and 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 5 | 5 | 7
score on a scale
  Baseline (Day 1) | 4.20 (3.83) | 6.20 (1.30) | 6.86 (4.53)
  Change from Baseline at Day 14: number analyzed (Participants) | 5 | 5 | 6
  Change from Baseline at Day 14 | -1.00 (2.92) | -0.40 (3.36) | -1.00 (2.28)
  Change from Baseline at Day 42: number analyzed (Participants) | 5 | 4 | 5
  Change from Baseline at Day 42 | -1.40 (2.70) | -2.00 (2.16) | 1.00 (2.92)
  Change from Baseline at Day 63: number analyzed (Participants) | 2 | 2 | 2
  Change from Baseline at Day 63 | -1.00 (1.41) | -2.50 (0.71) | -2.00 (1.41)
  Change from Baseline at Day 84: number analyzed (Participants) | 5 | 4 | 4
  Change from Baseline at Day 84 | 1.40 (4.51) | -1.25 (4.19) | -1.50 (1.29)

9. Secondary Outcome: Number of Participants With Daytime Sleepiness Assessed Using Sudden Onset of Sleep Questionnaire
Description: A sleep questionnaire was developed specifically for this study. Each participant (or support person for adolescents aged 15 to 17 years and for low-functioning participants) was asked to answer a series of 8 questions. The questions and their corresponding responses are as follows: a. Have you ever fallen asleep or have you been likely to fall asleep during your waking time? (Yes/No); b. Was this episode? (Gradual with awareness/Sudden and unpredictable/Sudden with awareness); c. Of the recent episode, how often does this occur? (Every day/Less frequently/Once a week/Other); d. Do you feel worried about falling asleep during the day? (Yes/No); e. Did the episode (or episodes) disrupt your daily activities? (Considerably/Marginally/No); f. Did this episode (or episodes) disrupt your social life (Considerably/Marginally/No); g. In the case of such an episode, was awakening? (Difficult/Easy/Normal). Categories with non-zero values are only reported here.
Time Frame: Baseline (Day 1), Days 7, 14, 42, 63, and 84
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 34 | 34 | 36
Participants
  a. Baseline: Day 1 (No): number analyzed (Participants) | 33 | 34 | 36
  a. Baseline: Day 1 (No) | 22 | 28 | 29
  a. Baseline: Day 1 (Yes): number analyzed (Participants) | 33 | 34 | 36
  a. Baseline: Day 1 (Yes) | 11 | 6 | 7
  a. Day 7 (No): number analyzed (Participants) | 31 | 33 | 32
  a. Day 7 (No) | 30 | 25 | 30
  a. Day 7 (Yes): number analyzed (Participants) | 31 | 33 | 32
  a. Day 7 (Yes) | 1 | 8 | 2
  a. Day 14 (No): number analyzed (Participants) | 30 | 32 | 34
  a. Day 14 (No) | 22 | 26 | 26
  a. Day 14 (Yes): number analyzed (Participants) | 30 | 32 | 34
  a. Day 14 (Yes) | 8 | 6 | 8
  a. Day 42 (No): number analyzed (Participants) | 32 | 32 | 32
  a. Day 42 (No) | 26 | 29 | 28
  a. Day 42 (Yes): number analyzed (Participants) | 32 | 32 | 32
  a. Day 42 (Yes) | 6 | 3 | 4
  a. Day 63 (No): number analyzed (Participants) | 3 | 2 | 2
  a. Day 63 (No) | 3 | 2 | 1
  a. Day 63 (Yes): number analyzed (Participants) | 3 | 2 | 2
  a. Day 63 (Yes) | 0 | 0 | 1
  a. Day 84 (No): number analyzed (Participants) | 33 | 31 | 31
  a. Day 84 (No) | 26 | 30 | 27
  a. Day 84 (Yes): number analyzed (Participants) | 33 | 31 | 31
  a. Day 84 (Yes) | 7 | 1 | 4
  b. Baseline: Day 1 (Gradual with Awareness): number analyzed (Participants) | 12 | 6 | 7
  b. Baseline: Day 1 (Gradual with Awareness) | 10 | 5 | 6
  b. Baseline: Day 1 (Sudden and Unpredictable (Without Awareness)): number analyzed (Participants) | 12 | 6 | 7
  b. Baseline: Day 1 (Sudden and Unpredictable (Without Awareness)) | 1 | 0 | 0
  b. Baseline: Day 1 (Sudden with Awareness): number analyzed (Participants) | 12 | 6 | 7
  b. Baseline: Day 1 (Sudden with Awareness) | 1 | 1 | 1
  b. Day 7 (Gradual with Awareness): number analyzed (Participants) | 1 | 8 | 2
  b. Day 7 (Gradual with Awareness) | 1 | 7 | 1
  b. Day 7 (Sudden and Unpredictable (Without Awareness)): number analyzed (Participants) | 1 | 8 | 2
  b. Day 7 (Sudden and Unpredictable (Without Awareness)) | 0 | 1 | 0
  b. Day 7 (Sudden with Awareness): number analyzed (Participants) | 1 | 8 | 2
  b. Day 7 (Sudden with Awareness) | 0 | 0 | 1
  b. Day 14 (Gradual with Awareness): number analyzed (Participants) | 10 | 7 | 8
  b. Day 14 (Gradual with Awareness) | 10 | 5 | 5
  b. Day 14 (Sudden and Unpredictable (Without Awareness)): number analyzed (Participants) | 10 | 7 | 8
  b. Day 14 (Sudden and Unpredictable (Without Awareness)) | 0 | 2 | 0
  b. Day 14 (Sudden with Awareness): number analyzed (Participants) | 10 | 7 | 8
  b. Day 14 (Sudden with Awareness) | 0 | 0 | 3
  b. Day 42 (Gradual with Awareness): number analyzed (Participants) | 7 | 3 | 4
  b. Day 42 (Gradual with Awareness) | 6 | 3 | 2
  b. Day 42 (Sudden with Awareness): number analyzed (Participants) | 7 | 3 | 4
  b. Day 42 (Sudden with Awareness) | 1 | 0 | 2
  b. Day 63 (Gradual with Awareness): number analyzed (Participants) | 1 | 0 | 1
  b. Day 63 (Gradual with Awareness) | 1 |  | 0
  b. Day 63 (Sudden with Awareness): number analyzed (Participants) | 1 | 0 | 1
  b. Day 63 (Sudden with Awareness) | 0 |  | 1
  b. Day 84 (Gradual with Awareness): number analyzed (Participants) | 7 | 1 | 5
  b. Day 84 (Gradual with Awareness) | 7 | 1 | 3
  b. Day 84 (Sudden and Unpredictable (Without Awareness)): number analyzed (Participants) | 7 | 1 | 5
  b. Day 84 (Sudden and Unpredictable (Without Awareness)) | 0 | 0 | 1
  b. Day 84 (Sudden with Awareness): number analyzed (Participants) | 7 | 1 | 5
  b. Day 84 (Sudden with Awareness) | 0 | 0 | 1
  c. Baseline: Day 1 (Everyday): number analyzed (Participants) | 10 | 6 | 7
  c. Baseline: Day 1 (Everyday) | 5 | 1 | 1
  c. Baseline: Day 1 (Less Frequently): number analyzed (Participants) | 10 | 6 | 7
  c. Baseline: Day 1 (Less Frequently) | 1 | 1 | 2
  c. Baseline: Day 1 (Once a Week): number analyzed (Participants) | 10 | 6 | 7
  c. Baseline: Day 1 (Once a Week) | 4 | 4 | 3
  c. Baseline: Day 1 (Other): number analyzed (Participants) | 10 | 6 | 7
  c. Baseline: Day 1 (Other) | 0 | 0 | 1
  c. Day 7 (Everyday): number analyzed (Participants) | 1 | 8 | 2
  c. Day 7 (Everyday) | 0 | 0 | 1
  c. Day 7 (Less Frequently): number analyzed (Participants) | 1 | 8 | 2
  c. Day 7 (Less Frequently) | 0 | 2 | 1
  c. Day 7 (Once a Month): number analyzed (Participants) | 1 | 8 | 2
  c. Day 7 (Once a Month) | 0 | 1 | 0
  c. Day 7 (Once a Week): number analyzed (Participants) | 1 | 8 | 2
  c. Day 7 (Once a Week) | 1 | 1 | 0
  c. Day 7 (Other): number analyzed (Participants) | 1 | 8 | 2
  c. Day 7 (Other) | 0 | 4 | 0
  c. Day 14 (Everyday): number analyzed (Participants) | 10 | 7 | 8
  c. Day 14 (Everyday) | 2 | 0 | 4
  c. Day 14 (Less Frequently): number analyzed (Participants) | 10 | 7 | 8
  c. Day 14 (Less Frequently) | 0 | 3 | 0
  c. Day 14 (Once a Week): number analyzed (Participants) | 10 | 7 | 8
  c. Day 14 (Once a Week) | 6 | 2 | 2
  c. Day 14 (Other): number analyzed (Participants) | 10 | 7 | 8
  c. Day 14 (Other) | 2 | 2 | 2
  c. Day 42 (Everyday): number analyzed (Participants) | 6 | 3 | 4
  c. Day 42 (Everyday) | 3 | 0 | 2
  c. Day 42 (Less Frequently): number analyzed (Participants) | 6 | 3 | 4
  c. Day 42 (Less Frequently) | 1 | 0 | 2
  c. Day 42 (Once a Month): number analyzed (Participants) | 6 | 3 | 4
  c. Day 42 (Once a Month) | 0 | 1 | 0
  c. Day 42 (Once a Week): number analyzed (Participants) | 6 | 3 | 4
  c. Day 42 (Once a Week) | 1 | 2 | 0
  c. Day 42 (Other): number analyzed (Participants) | 6 | 3 | 4
  c. Day 42 (Other) | 1 | 0 | 0
  c. Day 63 (Everyday): number analyzed (Participants) | 1 | 0 | 1
  c. Day 63 (Everyday) | 1 |  | 1
  c. Day 84 (Everyday): number analyzed (Participants) | 7 | 1 | 4
  c. Day 84 (Everyday) | 0 | 0 | 2
  c. Day 84 (Less Frequently): number analyzed (Participants) | 7 | 1 | 4
  c. Day 84 (Less Frequently) | 3 | 0 | 0
  c. Day 84 (Once a Week): number analyzed (Participants) | 7 | 1 | 4
  c. Day 84 (Once a Week) | 1 | 1 | 2
  c. Day 84 (Other): number analyzed (Participants) | 7 | 1 | 4
  c. Day 84 (Other) | 3 | 0 | 0
  d. Baseline: Day 1 (No): number analyzed (Participants) | 12 | 7 | 7
  d. Baseline: Day 1 (No) | 5 | 3 | 7
  d. Baseline: Day 1 (Yes): number analyzed (Participants) | 12 | 7 | 7
  d. Baseline: Day 1 (Yes) | 7 | 4 | 0
  d. Day 7 (No): number analyzed (Participants) | 1 | 8 | 2
  d. Day 7 (No) | 0 | 6 | 2
  d. Day 7 (Yes): number analyzed (Participants) | 1 | 8 | 2
  d. Day 7 (Yes) | 1 | 2 | 0
  d. Day 14 (No): number analyzed (Participants) | 10 | 7 | 8
  d. Day 14 (No) | 8 | 6 | 8
  d. Day 14 (Yes): number analyzed (Participants) | 10 | 7 | 8
  d. Day 14 (Yes) | 2 | 1 | 0
  d. Day 42 (No): number analyzed (Participants) | 6 | 3 | 4
  d. Day 42 (No) | 4 | 1 | 3
  d. Day 42 (Yes): number analyzed (Participants) | 6 | 3 | 4
  d. Day 42 (Yes) | 2 | 2 | 1
  d. Day 63 (No): number analyzed (Participants) | 1 | 0 | 1
  d. Day 63 (No) | 0 |  | 1
  d. Day 63 (Yes): number analyzed (Participants) | 34 | 0 | 1
  d. Day 63 (Yes) | 1 |  | 0
  d. Day 84 (No): number analyzed (Participants) | 7 | 1 | 4
  d. Day 84 (No) | 4 | 0 | 4
  d. Day 84 (Yes): number analyzed (Participants) | 7 | 1 | 4
  d. Day 84 (Yes) | 3 | 1 | 0
  e. Baseline: Day 1 (Considerably): number analyzed (Participants) | 12 | 7 | 7
  e. Baseline: Day 1 (Considerably) | 0 | 1 | 0
  e. Baseline: Day 1 (Marginally): number analyzed (Participants) | 12 | 7 | 7
  e. Baseline: Day 1 (Marginally) | 8 | 5 | 1
  e. Baseline: Day 1 (No): number analyzed (Participants) | 12 | 7 | 7
  e. Baseline: Day 1 (No) | 4 | 1 | 6
  e. Day 7 (Considerably): number analyzed (Participants) | 1 | 8 | 2
  e. Day 7 (Considerably) | 0 | 1 | 1
  e. Day 7 (Marginally): number analyzed (Participants) | 1 | 8 | 2
  e. Day 7 (Marginally) | 1 | 1 | 0
  e. Day 7 (No): number analyzed (Participants) | 1 | 8 | 2
  e. Day 7 (No) | 0 | 6 | 1
  e. Day 14 (Considerably): number analyzed (Participants) | 10 | 7 | 8
  e. Day 14 (Considerably) | 0 | 1 | 1
  e. Day 14 (Marginally): number analyzed (Participants) | 10 | 7 | 8
  e. Day 14 (Marginally) | 3 | 1 | 2
  e. Day 14 (No): number analyzed (Participants) | 10 | 7 | 8
  e. Day 14 (No) | 7 | 5 | 5
  e. Day 42 (Marginally): number analyzed (Participants) | 6 | 3 | 4
  e. Day 42 (Marginally) | 1 | 0 | 0
  e. Day 42 (No): number analyzed (Participants) | 6 | 3 | 4
  e. Day 42 (No) | 5 | 3 | 4
  e. Day 63 (Marginally): number analyzed (Participants) | 1 | 0 | 1
  e. Day 63 (Marginally) | 1 |  | 0
  e. Day 63 (No): number analyzed (Participants) | 1 | 0 | 1
  e. Day 63 (No) | 0 |  | 1
  e. Day 84 (Considerably): number analyzed (Participants) | 7 | 1 | 4
  e. Day 84 (Considerably) | 0 | 0 | 1
  e. Day 84 (Marginally): number analyzed (Participants) | 7 | 1 | 4
  e. Day 84 (Marginally) | 2 | 0 | 1
  e. Day 84 (No): number analyzed (Participants) | 7 | 1 | 4
  e. Day 84 (No) | 5 | 1 | 2
  f. Baseline: Day 1 (Marginally): number analyzed (Participants) | 12 | 7 | 7
  f. Baseline: Day 1 (Marginally) | 3 | 3 | 1
  f. Baseline: Day 1 (No): number analyzed (Participants) | 12 | 7 | 7
  f. Baseline: Day 1 (No) | 9 | 4 | 6
  f. Day 7 (Considerably): number analyzed (Participants) | 1 | 8 | 2
  f. Day 7 (Considerably) | 0 | 0 | 1
  f. Day 7 (Marginally): number analyzed (Participants) | 1 | 8 | 2
  f. Day 7 (Marginally) | 0 | 1 | 0
  f. Day 7 (No): number analyzed (Participants) | 1 | 8 | 2
  f. Day 7 (No) | 1 | 7 | 1
  f. Day 14 (Considerably): number analyzed (Participants) | 10 | 7 | 8
  f. Day 14 (Considerably) | 1 | 0 | 2
  f. Day 14 (Marginally): number analyzed (Participants) | 10 | 7 | 8
  f. Day 14 (Marginally) | 0 | 1 | 1
  f. Day 14 (No): number analyzed (Participants) | 10 | 7 | 8
  f. Day 14 (No) | 9 | 6 | 5
  f. Day 42 (Considerably): number analyzed (Participants) | 6 | 3 | 4
  f. Day 42 (Considerably) | 0 | 0 | 1
  f. Day 42 (Marginally): number analyzed (Participants) | 6 | 3 | 4
  f. Day 42 (Marginally) | 0 | 0 | 1
  f. Day 42 (No): number analyzed (Participants) | 6 | 3 | 4
  f. Day 42 (No) | 6 | 3 | 2
  f. Day 63 (No): number analyzed (Participants) | 1 | 0 | 1
  f. Day 63 (No) | 1 |  | 1
  f. Day 84 (Considerably): number analyzed (Participants) | 7 | 1 | 4
  f. Day 84 (Considerably) | 0 | 0 | 1
  f. Day 84 (Marginally): number analyzed (Participants) | 7 | 1 | 4
  f. Day 84 (Marginally) | 1 | 0 | 0
  f. Day 84 (No): number analyzed (Participants) | 7 | 1 | 4
  f. Day 84 (No) | 6 | 1 | 3
  g. Baseline: Day 1 (Difficult): number analyzed (Participants) | 12 | 7 | 7
  g. Baseline: Day 1 (Difficult) | 1 | 0 | 0
  g. Baseline: Day 1 (Easy): number analyzed (Participants) | 12 | 7 | 7
  g. Baseline: Day 1 (Easy) | 7 | 5 | 4
  g. Baseline: Day 1 (Normal): number analyzed (Participants) | 12 | 7 | 7
  g. Baseline: Day 1 (Normal) | 4 | 2 | 3
  g. Day 7 (Easy): number analyzed (Participants) | 1 | 8 | 2
  g. Day 7 (Easy) | 1 | 5 | 1
  g. Day 7 (Normal): number analyzed (Participants) | 1 | 8 | 2
  g. Day 7 (Normal) | 0 | 3 | 1
  g. Day 14 (Easy): number analyzed (Participants) | 10 | 7 | 8
  g. Day 14 (Easy) | 6 | 5 | 3
  g. Day 14 (Normal): number analyzed (Participants) | 10 | 7 | 8
  g. Day 14 (Normal) | 4 | 2 | 5
  g. Day 42 (Easy): number analyzed (Participants) | 6 | 3 | 4
  g. Day 42 (Easy) | 4 | 3 | 3
  g. Day 42 (Normal): number analyzed (Participants) | 6 | 3 | 4
  g. Day 42 (Normal) | 2 | 0 | 1
  g. Day 63 (Easy): number analyzed (Participants) | 1 | 0 | 1
  g. Day 63 (Easy) | 1 |  | 0
  g. Day 63 (Normal): number analyzed (Participants) | 1 | 0 | 1
  g. Day 63 (Normal) | 0 |  | 1
  g. Day 84 (Easy): number analyzed (Participants) | 7 | 1 | 4
  g. Day 84 (Easy) | 6 | 1 | 2
  g. Day 84 (Normal): number analyzed (Participants) | 7 | 1 | 4
  g. Day 84 (Normal) | 1 | 0 | 2

10. Secondary Outcome: Change From Baseline to Week 12 in Behavior/Symptoms as Measured by All Domains of the Repetitive Behavior Scale-Revised (RBS-R) Score
Description: The RBS-R is a 43-item informant-based questionnaire, assessing the variety of restricted and repetitive behaviors (RRBs) in individuals with ASD. The scale is grouped into six subscales: Stereotyped, Self-Injurious, Compulsive, Ritualistic, Sameness, and Restricted Behaviors. For each item, behaviors are rated on a 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. A total RBS-R score is calculated as the sum of the scores for the 43 items. The total score ranges from 0 to 129 and higher scores are indicative of more severe RRBs.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (80% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 30 | 29 | 28
score on a scale | -6.695 [-9.772 to -3.618] | -4.954 [-8.071 to -1.836] | -8.410 [-11.621 to -5.200]
Statistical Analysis 1: Comparison: Placebo vs Alogabat 20 mg; Test type: Superiority; p = 0.6082, ANCOVA; Difference in Adjusted Mean = 1.741, 80% CI 2-sided [-2.631 to 6.114]
Statistical Analysis 2: Comparison: Placebo vs Alogabat 60 mg; Test type: Superiority; p = 0.6228, ANCOVA; Difference in Adjusted Mean = -1.715, 80% CI 2-sided [-6.204 to 2.774]

11. Secondary Outcome: Change From Baseline to Week 12 on the Vineland-3 Socialization Domain
Description: Vineland-3 is a semi-structured interview measuring an individual's adaptive behavior across 3 domains: Communication, Socialization & Daily Living skills. Each domain consists of 3 subdomains. Subdomain raw scores are based on item responses (3-point scale: 0=never present; 1=sometimes present; 2=usually present) & are calculated for each subdomain of Socialization (interpersonal relationships, play and leisure time, coping skills) domain as sum of the scores for each item in the subdomain. Raw scores for the 3 Socialization subdomains are used to derive GSVs (range=10-164). A conversion table for mapping raw scores to GSV scores is found in the Vineland-3 manual (Sparrow et al. 2016). GSV is a person-ability score used to track an individual's progress. Vineland-3 Socialization Domain GSV score is calculated as a mean GSV score (summing the 3 GSV subdomain scores & dividing by 3). Vineland-3 Socialization Domain GSV score range = 10-145. Higher score =better adaptive functioning.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (80% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 31 | 27 | 29
score on a scale | 6.298 [4.302 to 8.294] | 3.315 [1.162 to 5.468] | 1.824 [-0.220 to 3.868]
Statistical Analysis 1: Comparison: Placebo vs Alogabat 20 mg; Test type: Superiority; p = 0.1987, ANCOVA; Difference in Adjusted Mean = -2.983, 80% CI 2-sided [-5.957 to -0.009]
Statistical Analysis 2: Comparison: Placebo vs Alogabat 60 mg; Test type: Superiority; p = 0.0460, ANCOVA; Difference in Adjusted Mean = -4.474, 80% CI 2-sided [-7.326 to -1.622]

12. Secondary Outcome: Change From Baseline to Week 12 on the Vineland-3 Communication Domain
Description: Vineland-3 is a semi-structured interview measuring an individual's adaptive behavior across 3 domains: Communication, Socialization & Daily Living skills. Each domain consists of 3 subdomains. Subdomain raw scores are based on item responses (3-point scale: 0=never present; 1=sometimes present; 2=usually present) & is calculated for each subdomain of the Communication (receptive, expressive, written) domain as the sum of the scores for each item within the subdomain. Raw scores for each of the 3 Communication subdomains are used to derive Growth Scale Values (GSVs; range from 10-197). A conversion table for mapping raw scores to GSV scores is found in Vineland-3 manual (Sparrow et al. 2016). GSV is a person-ability score used to track an individual's progress. Vineland-3 Socialization Domain GSV score is calculated as mean GSV score (summing the 3 GSV subdomain scores & dividing by 3). Vineland-3 Socialization Domain GSV score range=10-174. Higher score=better adaptive functioning.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (80% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
Number analyzed (Participants) | 32 | 27 | 28
score on a scale | 1.624 [0.087 to 3.162] | 2.903 [1.228 to 4.578] | 4.321 [2.693 to 5.948]
Statistical Analysis 1: Comparison: Placebo vs Alogabat 20 mg; Test type: Superiority; p = 0.4746, ANCOVA; Difference in Adjusted Means = 1.279, 80% CI 2-sided [-1.021 to 3.578]
Statistical Analysis 2: Comparison: Placebo vs Alogabat 60 mg; Test type: Superiority; p = 0.1244, ANCOVA; Difference in Adjusted Means = 2.697, 80% CI 2-sided [0.453 to 4.940]

ADVERSE EVENTS:
Time Frame: Up to Week 18
Description: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | Placebo | Alogabat 20 mg | Alogabat 60 mg
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 16/34 | 20/34 | 17/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | Alogabat 20 mg (N=34) | Alogabat 60 mg (N=36)
Fatigue (General disorders) | 0 (0) | 2 (5) | 3 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (7) | 3 (7) | 2 (12)
Hypersomnia (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (8) | 7 (7) | 6 (12)
Sudden onset of sleep (Nervous system disorders) | 0 (0) | 3 (6) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 2 (3) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT04299464/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04299464/SAP_001.pdf